CLINICAL TRIAL: NCT01460095
Title: Improving Access to HbA1c Measurement in Sub-Saharan Africa
Brief Title: Improving Access to HbA1c in Sub Saharan Africa
Acronym: IA3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yaounde Central Hospital (Other Government)
Collaborators: Newcastle University (Other); University of Yaounde 1 (Other)
Responsible Party: Principal Investigator, Sobngwi Eugene, Senior Lecturer and Consultant Physician, Yaounde Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: LT07-135
Record Dates: First submitted 2011-10-23; First posted 2011-10-26 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes Mellitus
Keywords: diabetes; translational research; HbA1c; education
MeSH Terms: conditions — Diabetes Mellitus | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HbA1c measurement and education (Experimental): 3-monthly Hba1c determination with immediate feedback and targeted education delivered to all participants
  Interventions: Other: HbA1c measurement and education

INTERVENTIONS:
Other: HbA1c measurement and education — three-monthly point of care measurement of HbA1c with immediate feedback to patients and provision of interpretation and targeted one-to-one education

SUMMARY:
Glycated haemoglobin (HbA1c) is the best surrogate of average blood glucose control in diabetic patients. Large-scale studies in the USA and UK have demonstrated that lowering HbA1c significantly reduces diabetes complications. Moreover, immediate feedback of HbA1c measurement to patients improves control. However, HbA1c is unavailable in most parts of Africa, a continent with one of the highest burden of diabetes. To translate these evidences, the investigators will provide affordable access to HbA1c measurement and relevant education in 2 African countries aiming significant improvement of diabetes control. The investigators will develop with local health authorities, training and cost-recovery scheme for long-term sustainability.

DETAILED DESCRIPTION:
The objective is to determine whether the introduction of routine affordable HbA1c determination with immediate feedback to patients and relevant education in an underserved population without any further intervention on drug supply would significantly improve diabetes control. As this will be an after-versus-before type study, each patient will be his own control.

Study setting The study will be undertaken in 10 existing diabetes care centre in two countries, including 4 regional centers in Guinea, a West African country of 10 millions inhabitants, and 6 regional centers in Cameroon, a Central African country of 18 million inhabitants.

The health districts covered in Guinea are Conakry, Labe, Kankan and Boke each being situated in a different ecological and cultural areas. In Cameroon, the health districts covered are Biyem Assi in Yaoundé, Garoua, Limbe, Ebolowa, Bamenda, Bafoussam also covering the 4 ecological zone of Cameroon.

All these health districts have existing diabetes care centre with trained personnel run in public hospital with prices and medicine affordable to most of the population covered. However, none of these centers have an HbA1c machine, and diabetes control is mainly evaluated using blood glucose, most often fasting.

Target population The aim is to provide the service to all patients followed in the selected centers at low cost however the first eligible 1000 patients will be included in the formal intervention free of charge.

Eligibility All patients with a physician-confirmed diagnosis of diabetes and who have been followed in the diabetes centre for at least one year are eligible Sample size In order to detect a difference of 1 unit (1% glycated haemoglobin) between to samples with a standard deviation of 1.2%, alpha coefficient of 0.001 and 0.8 power using a two-sided test, a minimum population of 80 subjects is required. The minimum sample size if alpha is 0.01 is 55 subjects. We therefore decided a sample size of 100 patients per centre in order to be able to analyze data taking into account center or physician effect. It thus give an overall sample size of 1000 subjects.

Sampling method We will use a systematic sampling, enrolling consecutive eligible patients volunteering to participate until completion of the sample size in each individual centre.

Inclusion All eligible patients, not intending to migrate from the study site within 1 year, and volunteering to participate will be enrolled. At inclusion the following will record of demographic characteristics, past medical history, characteristics of diabetes, evaluation of patient knowledge, and measurement of anthropometric characteristics, blood pressure, haematocrit, HbA1c, and urinary albumin excretion at baseline.

Intervention and follow up:

Data will be collected using a clinical record form designated to this effect. The intervention will consist of the measurement of HbA1c at baseline, 3, and 6 months with immediate feedback to patients and provision of targeted education after each determination, on level, significance, and targets.

Treatment will follow usual guidelines with no additional intervention. Adjustment of treatment will be done by the health care personnel in a treat-to-target fashion. No change in drug supply will be introduced. No specific recommendation will be given concerning the frequency of hospital visit between the study visits at baseline, month 3, 6, and 12. Each centre will continue with usual follow up frequency.

At month 12, we will repeat the evaluation of patient knowledge, and the measurement of anthropometric characteristics, blood pressure, haematocrit, HbA1c, and urinary albumin excretion for comparison to baseline.

Timeframe

* Start date: Month 7
* End of enrollment: Month 12
* End of follow-up of last patient enrolled: Month 24

Outcome measures

Primary outcome: Change in HbA1c from baseline to 12 months

Secondary outcomes:

* Change in percentage of patients at HbA1c target from baseline to 12 months
* Change in urinary albumin excretion from baseline to 12 months The other measures will serve for the interpretation of data Deliverables
* Dataset for each centre between Month 24 and Month 26

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diabetes mellitus irrespective of type
* Patients who have been followed regularly for at least one year prior to inclusion in the target health facilities
* Adult age (18 years and over)

Exclusion Criteria:

* Individuals planning to migrate from study sites within one year
* Any intercurrent acute illness
* Enrollment in any other concomitant intervention study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1349 (Actual)
Dates: Start 2009-03; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
one year change in glycated haemoglobin (HbA1c) | Baseline and 12 months
  Baseline to 12 months individual change in HbA1c level

SECONDARY OUTCOMES:
One-year change in proportion of patients reaching HbA1c targets | Baseline and 12 months
  Baseline to 12 months change in proportion of patients reaching HbA1c targets in each participating centre and in the overall population
One-year change in urinary albumin excretion | Baseline and 12 months
  Baseline to 12 months individual change in early morning sample urinary albumin excretion

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Sobngwi, MD, PhD, Principal Investigator — Newcastle University, UK and Yaounde Central Hospital, Cameroon
Locations (9):
- Cameroon (5):
  - Yaounde Central Hospital, Yaoundé, Centre Region
  - Garoua Regional Hospital, Garoua, North Region
  - Bamenda Regional Hospital, Bamenda, North-West Region
  - Buea Regional Hospital, Buea, South-West Region
  - Bafoussam District Hospital, Bafoussam
- Guinea (4):
  - Boke Regional Hospital, Boké
  - CHU Donka, Conakry
  - Kankan Regional Hospital, Kankan
  - Labe regional Hospital, Labé